CLINICAL TRIAL: NCT02656225
Title: Effect of Ejiao Compound in the Treatment of Postpartum Anemia of Qi-blood Deficiency Syndrome: Study Protocol of a Randomized Controlled Trial
Brief Title: Effect of Ejiao Compound in the Treatment of Postpartum Anemia of Qi-blood Deficiency Syndrome
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanfang Li, Associate chief physician, The First Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PA-1
Record Dates: First submitted 2015-12-31; First posted 2016-01-14 (Estimated); Last update posted 2016-03-29 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Anemia
Keywords: postpartum anemia; hemoglobin; iron metabolism; Traditional Chinese Medicine; Ejiao
MeSH Terms: interventions — Niferex

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ejiao compound (Experimental): The participants in experimental group receive Ejiao compound (20ml, twice daily) orally for 4 weeks.
  Interventions: Drug: Ejiao compound
- Niferex (Active Comparator): The participants in control group receive Polysaccharide Iron Complex(Niferex)(150mg per tablet, once daily) orally after breakfast over 4 weeks.
  Interventions: Drug: Niferex

INTERVENTIONS:
Drug: Ejiao compound — 20ml,twice daily, orally after breakfast Duration:4 weeks
  Other Names: Chinese patent medicine
  Arms: Ejiao compound
Drug: Niferex — one tablet,once daily, orally after breakfast Duration:4 weeks
  Other Names: Polysaccharide Iron Complex
  Arms: Niferex

SUMMARY:
The prevalence of postpartum anemia is a great threat for maternal and infant health without timely and effective treatment. Oral iron therapy has been used for centuries as a treatment of anemia, however, it is noteworthy that treatment with oral iron might have a limited, and even a harmful role in some clinical scenarios. Ejiao compound is composed with donkey-hide glue, Ginseng, Codonopsis pilosula, prepared rhizome of rehmannia, and crab apple, which has been widely used in the treatment of various types of anemia in China for decades and might be a potentially effective therapy for postpartum anemia. Recently, studies involving animal subjects have helped shed light on its mechanism of action.

In this study, the investigators aimed to conduct a randomized controlled trial to assess the efficacy and safety of Ejiao compound comparing with oral iron in the treatment of mild postpartum anemia with or without iron deficiency.

DETAILED DESCRIPTION:
1. Study type: This is a randomized, parallel controlled and single blind study. The sample ratio of the experimental group and the control group will be 1:1.
2. Study Setting and Recruitment: All participants experience vaginal delivery and are diagnosed with mild postpartum anemia. They will be recruited from the obstetric inpatient department in two hospitals: the first affiliated hospital of Guangzhou University of Traditional Chinese Medicine, and Maternal and Child Health Hospital of Panyu District in Guangzhou City. All assessments and interventions will occur at hospitals.
3. Randomization, blinded method, and allocation concealment: Patients meeting the criteria were randomized into experimental group or control group, according to a computer-generated list. The patients in experimental group will receive the treatment of Ejiao compound while the patients in control group will be treated by Polysaccharide iron complex. The study physicians will receive a sealed decoding envelope per treatment, they will not know the identity of the participants, will not handle the study products, will not know the assigned treatment, and will not share their own examination results. After receiving the evaluation by the study physicians and finishing the investigation form, the patient will take her own sealed decoding envelope and go to the pharmacy of the clinical trial center to receive her medication. The staff of the pharmacy of the clinical trial center is responsible for the distribution and return of experimental drugs to patients. All envelopes, sealed or unsealed, will be returned to the investigators at the end of the study. Patients would be required to return boxes whether they are used and unused at each visit and compliance will be assessed by counting the bottles and capsules.
4. Sample size calculation: It was reported that treatment with oral iron for anemia in postpartum women increase the Hb concentration by 49.3% by day 40. Combined with etiological treatment, Ejiao compound used to treat anemia in non pregnant population for three months, the Hb concentration increased by 66.9%. Basing on the results of literatures mentioned above, the investigators suppose that the difference of Hb concentration between patients only receiving the Ejiao compound for 4 weeks and patients only receiving oral iron for 4 weeks would be 25.0%. The α-value is set at 0.05 and the test power is 0.90. The final sample size should be 68 in each group. With an anticipated dropout rate of 20% during the follow-up, the initial sample size for each group should be 85, and 170 in total for two groups.
5. Statistical analysis: The statisticians will be blinded to the allocation of the participants. Statistics Package for Social Science (SPSS)19.0 statistical software packages will be used to analyze the data. The intention-to-treat population will include all randomized patients who receive the assigned treatment at least once, and who have an evaluation of outcomes. The measurement data will be analyzed by using t-test or the rank sum test, and the numeration data will be analyzed by using chi-square test or Fisher's exact test. P<0.05 indicates statistical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years to 45 years with mild postpartum anemia (Hb <10 g/dl and ≥7 g/dl at 24-48 hours postpartum);
2. Absence of antepartum anemia, which is defined as Hb≥11.0 g/dL within 48 hours before delivery;
3. Singleton pregnancy;
4. Type of syndrome in Traditional Chinese Medicine is "Qi-blood deficiency".
5. Patients having not received blood transfusion or any forms of anti-anemia treatment in Western medicine or TCM in the last 12 weeks;
6. Informed consent obtained.

Exclusion Criteria:

1. Type of syndrome in TCM is NOT "Qi-blood deficiency";
2. Antepartum anemia;
3. Twin or multiple pregnancies;
4. A history of haematological disease (e.g. sickle cell anemia or thalassemias);
5. A history of undigestive disease (e.g. gastric ulcer, gastritis) or inflammatory bowel disease;
6. A history of cardiovascular diseases, renal or liver disease, asthma, thromboembolism, HIV infection, tuberculosis, cancer and seizures;
7. Patients having received blood transfusion or any forms of anti-anemia treatment in Western medicine or TCM in the last 12 weeks;
8. Alcohol or drug abuse;
9. Patients with mental illness or poor compliance to medical treatment;
10. Participation in another clinical trial within the previous three months;
11. No informed consent obtained.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 170 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin(Hb) | before and after treatment

SECONDARY OUTCOMES:
Serum ferritin | before and after treatment
Life quality assessment: a Health Assessment Questionnaire(The Short Form-36 Health Survey, SF-36) | before and after treatment
Traditional Chinese Medicine symptom score:a self-made scale for Qi-blood Deficiency Syndrome | before and after treatment

OTHER OUTCOMES:
Adverse reactions or events: renal function | before and after treatment
  serum creatinine and urea nitrogen
Adverse reactions or events: liver function | before and after treatment
  aspartate aminotransferase(AST), alanine aminotransferase (ALT)

CONTACTS AND LOCATIONS:
Overall Officials: yanfang Li, PhD, Study Chair — the First Affiliated Hospital, Guangzhou University of Chinese Medicine
Locations (1):
- the First Affiliated Hospital, Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dodd J, Dare MR, Middleton P. Treatment for women with postpartum iron deficiency anaemia. Cochrane Database Syst Rev. 2004 Oct 18;2004(4):CD004222. doi: 10.1002/14651858.CD004222.pub2. PMID 15495089
- [Background] Bhandal N, Russell R. Intravenous versus oral iron therapy for postpartum anaemia. BJOG. 2006 Nov;113(11):1248-52. doi: 10.1111/j.1471-0528.2006.01062.x. Epub 2006 Sep 27. PMID 17004982
- [Background] Ramakers C, van der Woude DA, Verzijl JM, Pijnenborg JM, van Wijk EM. An added value for the hemoglobin content in reticulocytes (CHr) and the mean corpuscular volume (MCV) in the diagnosis of iron deficiency in postpartum anemic women. Int J Lab Hematol. 2012 Oct;34(5):510-6. doi: 10.1111/j.1751-553X.2012.01423.x. Epub 2012 May 1. PMID 22548729
- [Background] Breymann C, Honegger C, Holzgreve W, Surbek D. Diagnosis and treatment of iron-deficiency anaemia during pregnancy and postpartum. Arch Gynecol Obstet. 2010 Nov;282(5):577-80. doi: 10.1007/s00404-010-1532-z. Epub 2010 Jun 25. PMID 20577752
- [Background] Milman N. Postpartum anemia I: definition, prevalence, causes, and consequences. Ann Hematol. 2011 Nov;90(11):1247-53. doi: 10.1007/s00277-011-1279-z. Epub 2011 Jun 28. PMID 21710167
- [Background] Milman N. Postpartum anemia II: prevention and treatment. Ann Hematol. 2012 Feb;91(2):143-54. doi: 10.1007/s00277-011-1381-2. Epub 2011 Dec 9. PMID 22160256
- [Background] Bergmann RL, Richter R, Bergmann KE, Dudenhausen JW. Prevalence and risk factors for early postpartum anemia. Eur J Obstet Gynecol Reprod Biol. 2010 Jun;150(2):126-31. doi: 10.1016/j.ejogrb.2010.02.030. Epub 2010 Mar 29. PMID 20303210